CLINICAL TRIAL: NCT01391676
Title: Imaging of Blebs After Trabeculectomy With Mitomycin C 0,02% Using the Spectral Domain Optical Coherence Tomography
Brief Title: Imaging of Trabeculectomy Blebs Using the Spectral Domain Optical Coherence Tomography
Acronym: SDOCT-TE
Status: Completed | Type: Observational
Sponsor: Technische Universität Dresden (Other)
Responsible Party: Principal Investigator, Dr. Karin Pillunat, Principal Investigator, Technische Universität Dresden
Other Study IDs: SD OCT-TE
Record Dates: First submitted 2011-07-08; First posted 2011-07-12 (Estimated); Last update posted 2013-09-10 (Estimated); Status verified 2013-09

CONDITIONS: Glaucoma; Filtering Blebs
Keywords: glaucoma; trabeculectomy; filtering bleb; spectral domain optical coherence tomography
MeSH Terms: conditions — Glaucoma | interventions — Trabeculectomy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Trabeculectomy: glaucoma patients undergoing trabeculectomy with mitomycin c 0,02%
  Interventions: Procedure: trabeculectomy

INTERVENTIONS:
Procedure: trabeculectomy — postoperative imaging of trabeculectomy blebs with the spectral domain optical coherence tomography

SUMMARY:
The aim of this study is imaging of trabeculectomy blebs regarding structure and function with the spectral domain optical coherence tomography.

DETAILED DESCRIPTION:
After a trabeculectomy with mitomycin C 0,02% for 3 minutes, the blebs are controlled by a glaucoma specialist on day 1, week 1,2,3,4, month 3 and 6 after surgery. The glaucoma specialist will evaluate the bleb appearance according to a standardized protocol. At the same time points the bleb will be imaged with the spectral domain optical coherence tomography, to monitor bleb changes objectively. The investigators hope to see signs of bleb incapsulation and scarring earlier and then treat the patient accordingly.

ELIGIBILITY:
Inclusion Criteria:

glaucoma patients who need a trabeculectomy with mitomycin C 0,02% for further reduction of intraocular pressure, informed consent

Exclusion Criteria:

patient without glaucoma, under 18 years of age, not willing to take part in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: glaucoma patients who need a trabeculectomy with mitomycin C 0,02% for further reduction of intraocular pressure (IOP)
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2011-03; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
grading of filtering bleb | December 2011

CONTACTS AND LOCATIONS:
Overall Officials: Karin R Hornykewycz, MD, Principal Investigator — University Eye Clinic Dresden, Fetscherstrasse 74, 01307 Dresden, Germany
Locations (1):
- University Eye Clinic Dresden, Dresden, Saxony, Germany